CLINICAL TRIAL: NCT03640234
Title: Return of Actionable Variants Empirical (RAVE) Study
Brief Title: Return of Actionable Variants Empirical Study
Acronym: RAVE
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Principal Investigator, Iftikhar J. Kullo, Principal Investigator, Mayo Clinic
Other Study IDs: 15-005013; U01HG006379 (NIH)
Record Dates: First submitted 2018-07-23; First posted 2018-08-21 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA obtained from blood samples in the primary cohort and from saliva in family members.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a genomic implementation project with ancillary studies to understand the impact on patients' health and well-being of returning genomic results to them and depositing those results in the medical record.

DETAILED DESCRIPTION:
Study participant DNA samples will be sequenced for 109 genes of interest along with genotyping of select polymorphisms. Genetic tests will be performed in a Clinical Laboratory Improvement Amendments (CLIA) certified lab (Baylor Human Genome Sequencing Laboratory). Selected results (pathogenic/likely pathogenic) will be returned to participants by a genetic counselor and deposited into the Electronic Health Record (EHR).

ELIGIBILITY:
Inclusion Criteria:

* Moderate to Severe Hypercholesterolemia, elevated triglycerides, or colon polyps
* Resident of southeast Minnesota area
* Able to provide informed consent
* Current participant in the Mayo Clinic Biobank (08-007049, Cerhan PI), the Vascular Disease Biorepository (08-008355, Kullo PI), or the Study of the Genetic Determinants of Peripheral Artery Disease (PAD) (06-002911, Kullo PI) with blood derived DNA available

Exclusion Criteria:

* Pregnant women will be allowed to enroll in the study. This is not an interventional study and there will be no risk to the mother or neonate. Other vulnerable study populations will be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We recruited 3030 participants from Mayo Clinic biobanks in Rochester, MN, who had hypercholesterolemia, colon polyps or both, thereby enriching for FH.
Sampling Method: Non-Probability Sample
Enrollment: 418 (Actual)
Dates: Start 2016-02-25 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Participant utilization of clinical resources following the return of medically actionable genetic variants. | Feb 2016-June 2020
  The EHR of study participants will be periodically reviewed beginning 6 months following the disclosure of results. EHR documented utilization of clinical resources by participants (e.g. lipid profile for cholesterol measurement, mammogram, colonoscopy, prophylactic surgery, etc.) will be reviewed to assess whether the disclosure of actionable genetic findings led to initiation of medical therapy or ordering of additional tests. Data will be manually abstracted into condition-specific REDCap questionnaires which are harmonized across multiple eMERGE Network sites.

SECONDARY OUTCOMES:
The number of new cases detected as a result of cascade screening in the family members | Feb 2017- Dec 2020
  This outcome is being assessed as a supplemental study that includes patients with definite, probable and possible Familial Hypercholesterolemia (FH). We will compare the yield of cascade screening in FH patients with and without an identifiable pathogenic variant. We will enroll 50 patients with definite FH by recruiting an additional 25 from the FH Clinic at Mayo and 50 patients each with probable and possible FH, matching on age and sex. Family members of patients with definite FH will undergo testing for the relevant pathogenic variant using saliva kits and family members of those with probable/possible FH will have a lipid profile checked. We will assess the number of new cases detected (defined as presence of a pathogenic variant in the family member of definite FH patient or LDL-C >155 mg/dL (>130 mg/dL in children) in family members of probable/possible FH patients, and the cost of detecting a new case.
Total Expense due to disclosure of actionable variants | 4 years
  The EHR will be periodically reviewed after disclosure of results to assess whether the disclosure led to initiation of medical therapy or ordering of additional tests. Measured in U.S. dollars.
Participant intent-to-share genetic test results | Sept 2017-June 2020
  Participants are offered pre-and-post-counseling questionnaires, provide pedigree information, and family member contact information. Questionnaires include measures of intent-to-share and barriers to sharing genetic results.
Number of first-degree relatives per proband and number of contacted first-degree relatives per proband | Sept 2017-Dec 2020
  The number of first-degree relatives will be assessed using patient-provided family history information. The number of contacted family members will be assessed by measuring family member response to participant contact materials.
Family member uptake of genetic testing | Sept 2017- Dec 2020
  Family member respondents who provide consent will be offered genetic testing. The uptake of genetic testing will be documented for each family member.

REFERENCES:
- [Background] Kaphingst KA, McBride CM, Wade C, Alford SH, Reid R, Larson E, Baxevanis AD, Brody LC. Patients' understanding of and responses to multiplex genetic susceptibility test results. Genet Med. 2012 Jul;14(7):681-7. doi: 10.1038/gim.2012.22. PMID 22481132
- [Background] Brehaut JC, O'Connor AM, Wood TJ, Hack TF, Siminoff L, Gordon E, Feldman-Stewart D. Validation of a decision regret scale. Med Decis Making. 2003 Jul-Aug;23(4):281-92. doi: 10.1177/0272989X03256005. PMID 12926578
- [Background] Zick CD, Mathews CJ, Roberts JS, Cook-Deegan R, Pokorski RJ, Green RC. Genetic testing for Alzheimer's disease and its impact on insurance purchasing behavior. Health Aff (Millwood). 2005 Mar-Apr;24(2):483-90. doi: 10.1377/hlthaff.24.2.483. PMID 15757934
- [Background] Dunlay SM, Shah ND, Shi Q, Morlan B, VanHouten H, Long KH, Roger VL. Lifetime costs of medical care after heart failure diagnosis. Circ Cardiovasc Qual Outcomes. 2011 Jan 1;4(1):68-75. doi: 10.1161/CIRCOUTCOMES.110.957225. Epub 2010 Dec 7. PMID 21139091
- [Background] Lipscomb J, Ancukiewicz M, Parmigiani G, Hasselblad V, Samsa G, Matchar DB. Predicting the cost of illness: a comparison of alternative models applied to stroke. Med Decis Making. 1998 Apr-Jun;18(2 Suppl):S39-56. doi: 10.1177/0272989X98018002S07. PMID 9566466
- [Background] Gaff CL, Clarke AJ, Atkinson P, Sivell S, Elwyn G, Iredale R, Thornton H, Dundon J, Shaw C, Edwards A. Process and outcome in communication of genetic information within families: a systematic review. Eur J Hum Genet. 2007 Oct;15(10):999-1011. doi: 10.1038/sj.ejhg.5201883. Epub 2007 Jul 4. PMID 17609674
- [Background] Hughes C, Lerman C, Schwartz M, Peshkin BN, Wenzel L, Narod S, Corio C, Tercyak KP, Hanna D, Isaacs C, Main D. All in the family: evaluation of the process and content of sisters' communication about BRCA1 and BRCA2 genetic test results. Am J Med Genet. 2002 Jan 15;107(2):143-50. doi: 10.1002/ajmg.10110. PMID 11807889
- [Background] Talmud PJ, Drenos F, Shah S, Shah T, Palmen J, Verzilli C, Gaunt TR, Pallas J, Lovering R, Li K, Casas JP, Sofat R, Kumari M, Rodriguez S, Johnson T, Newhouse SJ, Dominiczak A, Samani NJ, Caulfield M, Sever P, Stanton A, Shields DC, Padmanabhan S, Melander O, Hastie C, Delles C, Ebrahim S, Marmot MG, Smith GD, Lawlor DA, Munroe PB, Day IN, Kivimaki M, Whittaker J, Humphries SE, Hingorani AD; ASCOT investigators; NORDIL investigators; BRIGHT Consortium. Gene-centric association signals for lipids and apolipoproteins identified via the HumanCVD BeadChip. Am J Hum Genet. 2009 Nov;85(5):628-42. doi: 10.1016/j.ajhg.2009.10.014. PMID 19913121
- [Background] Futema M, Shah S, Cooper JA, Li K, Whittall RA, Sharifi M, Goldberg O, Drogari E, Mollaki V, Wiegman A, Defesche J, D'Agostino MN, D'Angelo A, Rubba P, Fortunato G, Walus-Miarka M, Hegele RA, Aderayo Bamimore M, Durst R, Leitersdorf E, Mulder MT, Roeters van Lennep JE, Sijbrands EJ, Whittaker JC, Talmud PJ, Humphries SE. Refinement of variant selection for the LDL cholesterol genetic risk score in the diagnosis of the polygenic form of clinical familial hypercholesterolemia and replication in samples from 6 countries. Clin Chem. 2015 Jan;61(1):231-8. doi: 10.1373/clinchem.2014.231365. Epub 2014 Nov 20. PMID 25414277
- [Derived] Miller AA, Bangash H, Smith CY, Wood-Wentz CM, Bailey KR, Kullo IJ. A pragmatic clinical trial of cascade testing for familial hypercholesterolemia. Genet Med. 2022 Dec;24(12):2535-2543. doi: 10.1016/j.gim.2022.08.026. Epub 2022 Sep 29. PMID 36173399
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials